CLINICAL TRIAL: NCT05600998
Title: Exploratory Clinical Study of Camrelizumab in Combination With Anlotinib in the Treatment of Patients With Advanced Ovarian Clear Cell Carcinoma
Brief Title: A Study of Camrelizumab in Combination With Anlotinib in Subjects Advanced Ovarian Clear Cell Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-SHR1210
Record Dates: First submitted 2022-10-09; First posted 2022-11-01 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Ovarian Clear Cell Carcinoma
MeSH Terms: interventions — camrelizumab; anlotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab+Anlotinib (Experimental): Subjects will receive carilizumab every three weeks, with alozantinib 20 mg orally daily for 9 weeks
  Interventions: Drug: Camrelizumab

INTERVENTIONS:
Drug: Camrelizumab — Subjects will receive carilizumab every three weeks, with alozantinib 20 mg orally daily for 9 weeks
  Other Names: Anlotinib

SUMMARY:
This study is prospective ,open-label, single-center phase II clinical study. Target population is patients with advanced (stage III-IV) ovarian clear cell carcinoma. Study objective is to evaluate effectiveness response of Camrelizumab + anlotinib in subjects with advanced ovarian clear cell carcinoma Camrelizumab is a humanized anti-PD1 IgG4 monoclonal antibody.

DETAILED DESCRIPTION:
In this study, eligible subjects were given a combination of carrelizumab and alozantinib at the same time, repeated every 21 days, during treatment based on imaging evaluation of the patient if disease progression, toxicity intolerance, or other reasons specified by the regimen could be terminated.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years; 2. Pathohistological or cytology confirmed as ovarian transparent cell carcinoma, and FIGO stage in 2018 is stage III-IV; ≥ four courses of chemotherapy and failed to reach CR 3. ECOG score; 0-2 points; 4. Expected survival ≥ 3 months; 5. The investigator confirmed to have at least one measurable lesion (10 mm long diameter of CT scan of tumor lesions ≥10 mm, short diameter of CT scan of lymph node lesions ≥15 mm)) according to the RECIST 1.1 standard), or ascites 6. The main organs function normally, and the test results during screening must meet the following requirements:

1. Blood routine examination criteria should be met (no blood transfusion and blood products within 14 days, no use of G-CSF and other hematopoietic stimulating factors to correct):

   A. Hemoglobin (Hb) ≥ 80 g/L; B. Number of neutrophils (ANC) ≥ 1.5 × 109/L; C. Platelet count (PLT) ≥ 80 ×109/L;
2. Biochemical inspection must meet the following standards:

A. Total bilirubin (TBIL) < 1.5 Upper limit of normal value (ULN); B. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 2.5 ULL compared <with 5 ULN for patients with liver metastases; C. serum creatinine (Cr) ≤ 1.5 ULN or endogenous creatinine clearance > 60 ml/min (Cockcroft-Galt formula); D. Urine routine test results show urine protein (UPRO) < 2+ or 24-hour urine protein quantitative <1 g; 7. Women of gestational age must agree to adequate contraception for the entire duration of the study and within 6 months after the end of treatment.

8.Signed a written informed consent form with good expected adherence to the research protocol.

Exclusion Criteria:

1. Have previously received anti-PD-1, anti-PD-L1, anti-PD-L2, or anti-CTLA-4 antibodies (or any other antibodies acting on the T cell synergistic stimulation or checkpoint pathway);
2. Previous exposure to other anti-angiogenic small molecule TKI drugs, such as apatinib, alotinib, sorafinil, regofinib, etc.;
3. Patients with active brain metastases (for patients with stable symptoms after treatment of brain metastases, they can be selected if they remain in a stable state for at least 4 weeks);
4. Immunosuppressive drugs have been used within 28 days before the first use of carirelizumab, excluding nasal and inhaled corticosteroids or systemic steroid hormones in physiological doses (i.e., prednisolone or other corticosteroids of equivalent pharmacophysiological doses not exceeding 10 mg / day);
5. Received systematic systemic therapy with anti-tumor indications of Chinese herbal medicine or immunomodulatory effect (including thymus peptide, interferon, interleukin, except for the control of pleural effusion topical use) within 2 weeks before the first administration;
6. Suffering from serious cardiovascular diseases: myocardial ischemia or myocardial infarction above grade II, poorly controlled arrhythmias (including QTc interval men ≥ 450 ms, women ≥ 470 ms); Grade III. to IV. cardiac insufficiency (see Annex 3 according to the NYHA grade of the New York Cardiology Society), or if the left ventricular ejection fraction (LVEF) < 50% on cardiac color ultrasound;
7. Complicated by severe infection within 4 weeks before the first medication (eg, intravenous infusion of antibiotics, antifungal or antiviral drugs), or unexplained fever > during screening / before the first administration 38.5°C； or major surgical treatment within 3 weeks prior to the first medication;
8. The presence of active autoimmune diseases or immunodeficiency, or the history of the above, including but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, rheumatoid arthritis, inflammatory bowel disease, pituititis, vasculitis, nephritis, etc.) shall not be included. The following exceptions are those with a history of autoimmune hypothyroidism but receiving thyroid hormone replacement therapy. After treatment with an insulin dosing regimen, patients with type 1 diabetes whose blood glucose is controlled may participate in this study.
9. Subjects undergo systematic treatment such as bronchodilators, asthma control is not satisfactory, can not be included (asthma in childhood has been completely resolved, adults do not need any intervention can be included).
10. Human immunodeficiency virus (HIV) infection or known to have acquired immunodeficiency syndrome (AIDS), untreated active hepatitis B, hepatitis C (hepatitis C antibody positive, and HCV-RNA is higher than the lower limit of detection of analytical methods) or co-infection with hepatitis B and C;
11. The subject has received or plans to receive a transplant of a solid organ or blood system during the study (except for corneal transplantation);
12. Are currently participating in interventional clinical research or has been treated with other experimental drugs or research devices within 4 weeks prior to the first dose; Adequate recovery from toxicity and/or complications caused by any intervention before the first dose (i.e., ≦ grade 1 or at baseline, excluding fatigue or hair loss);
13. Have a clear history of allergies, may be potentially allergic or intolerant to the test drug and its similar biological agents;
14. Those with a history of psychotropic drug abuse and who cannot be withdrawn or have mental disorders;
15. People with a history of hereditary or acquired bleeding or coagulation dysfunction (it is up to the investigator to determine whether they can be selected)
16. Uncontrolled hypertension (systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥90 mmHg, despite optimal drug therapy);
17. Those who have had significant coughing up blood 2 months prior to entry into the study, or who have had a daily hemoptysis volume of half a teaspoon (2.5 ml) or more; or have had clinically significant bleeding symptoms or a clear tendency to bleed within 3 months prior to the study, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, or vasculitis; or arteriovenous thrombosis events that occurred within 6 months prior to the study, such as cerebrovascular accidents (including temporary ischemic attacks, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism;
18. Abnormal coagulation function (INR>1.5 or prothrombin time (PT)>ULN+4 seconds or APTT >1.5ULN), with bleeding tendencies or being undergoing thrombolytic or anticoagulant therapy;
19. Urine routine suggests that urine protein ≥++, or confirm that the amount of urine protein ≥ 1.0g in 24 hours;
20. Increases the risk associated with participating in a study or trial drug and, according to the investigator's judgment, can lead to other circumstances in which the patient is unsuitable for the study to be selected.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-10-30 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | 12 weeks
  Evaluated according to RECIST1.1, refers to the proportion of patients whose tumors shrink to a certain amount and remain for a certain period of time. Specifically, the proportion of the total number of treated CR+PR cases to the overall number of measurable cases.

SECONDARY OUTCOMES:
Progression-free survival | 12weeks
  Defined as the date on which the subject begins with the first treatment to the date on which the tumor progression is first recorded or dies for any reason, whichever appears first.

CONTACTS AND LOCATIONS:
Overall Officials: Hongyan Guo, Doctor, Principal Investigator — Peking University Third Hospital

IPD SHARING:
Plan to Share IPD: No